CLINICAL TRIAL: NCT04654572
Title: The Investigation of Muscle Mechanical Properties in Burned Patients.
Brief Title: The Mechanical Properties of Burned Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Assistant of professeur, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2018-05
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Burns; Muscle Loss; Viscoelastic Properties; Stiffness
Keywords: Burn; muscle; myotonometer; viscoelasticity; stiffness
MeSH Terms: conditions — Burns; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- burned group (Experimental): burned patients
  Interventions: Diagnostic Test: Myotonometric measurement
- control group (Experimental): sedentary people
  Interventions: Diagnostic Test: Myotonometric measurement

INTERVENTIONS:
Diagnostic Test: Myotonometric measurement — Myotonometric assessment can predict the muscle stiffness, tone and elasticity

SUMMARY:
The investigate of mechanical properties of muscles in burned patients.

DETAILED DESCRIPTION:
The hypermetabolic response to severe burn is characterized by muscle protein catabolism. Current opinion states that the hypermetabolic state resolves soon after complete wound closure. Clinically, we have witnessed that burned patient appear to be hypermetabolic and catabolic long after full healing of their wounds. Our goal in this study was to determine muscle mechanical properties (tone, stiffness and elasticity) after burn.

ELIGIBILITY:
Inclusion Criteria:

* burned patient
* major burn over %20 TBSA

Exclusion Criteria:

* Amputation
* Dead
* Systemic disease and abuse

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Stiffness | 6 week
  Myotonometric measurement was used to determine for muscle stiffness. Device has a probe that creates constant pre-excitations and generates short-term, low-force mechanical stimulations over skin. The stimulations induce damped natural oscillations in the tissue and the myoton device records these oscillations with an accelerometer. Muscle tone, elasticity, and stiffness are calculated separately by the device.
Elasticity | 6 week
  Myotonometric measurement was used to determine for muscle elasticity. Device has a probe that creates constant pre-excitations and generates short-term, low-force mechanical stimulations over skin. The stimulations induce damped natural oscillations in the tissue and the myoton device records these oscillations with an accelerometer. Muscle tone, elasticity, and stiffness are calculated separately by the device.
Tone | 6 week
  Myotonometric measurement was used to determine for muscle tone. Device has a probe that creates constant pre-excitations and generates short-term, low-force mechanical stimulations over skin. The stimulations induce damped natural oscillations in the tissue and the myoton device records these oscillations with an accelerometer. Muscle tone, elasticity, and stiffness are calculated separately by the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan kalyoncu üniversity, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data of myotonometric measurement and physical characteristics of participants will share
Supporting Information: Study Protocol, CSR
Time Frame: after publication and 10 years

REFERENCES:
- [Background] Gittings PM, Grisbrook TL, Edgar DW, Wood FM, Wand BM, O'Connell NE. Resistance training for rehabilitation after burn injury: A systematic literature review & meta-analysis. Burns. 2018 Jun;44(4):731-751. doi: 10.1016/j.burns.2017.08.009. Epub 2017 Oct 7. PMID 29017743
- [Background] Porter C, Hardee JP, Herndon DN, Suman OE. The role of exercise in the rehabilitation of patients with severe burns. Exerc Sport Sci Rev. 2015 Jan;43(1):34-40. doi: 10.1249/JES.0000000000000029. PMID 25390300
- [Background] Ianieri G, Saggini R, Marvulli R, Tondi G, Aprile A, Ranieri M, Benedetto G, Altini S, Lancioni GE, Goffredo L, Bellomo RG, Megna M, Megna G. New approach in the assessment of the tone, elasticity and the muscular resistance: nominal scales vs MYOTON. Int J Immunopathol Pharmacol. 2009 Jul-Sep;22(3 Suppl):21-4. doi: 10.1177/03946320090220S304. No abstract available. PMID 19887038